CLINICAL TRIAL: NCT06154642
Title: Physiological Study of Hemodynamic and Microcirculatory Evolution Before/After Transcatheter Aortic Valve Replacement (TAVI)
Brief Title: Perioperative Hemodynamic and Microcirculatory Physiological Study During TAVI
Acronym: TAVI
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Collaborators: Stanislas Abrard (Unknown); Noble Stéphane (Unknown)
Responsible Party: Principal Investigator, Karim Bendjelid, Prof., University Hospital, Geneva
Other Study IDs: 2023-01118
Record Dates: First submitted 2023-11-23; First posted 2023-12-04 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Aortic Valve Stenosis
Keywords: Transcatheter Aortic Valve Implantation; Microcirculation; Endothelium, vascular; Microvascular reactivity
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Echocardiography; Photoplethysmography; Perfusion Index; Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — ethylenediaminetetraacetic acid plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Determination of arterial compliance using blood pressure waveform analysis — Measurement of arterial stiffness using a non-invasive pressure transducer placed on the skin of the wrist, which records the pulse wave at the level of the radial artery in order to analyze the characteristics of the arterial wall. The parameters of interest are the arterial stiffness of large- and small-caliber arteries (ml/mmHg).
  Other Names: Arterial tonometry
Diagnostic Test: Measurement of plasma Vascular Endothelium Growth Factor — Measurement of plasma Vascular Endothelium Growth Factor levels by ELISA
  Other Names: Vascular Endothelium Growth Factor
Diagnostic Test: Skin temperature gradient — Measurement of skin surface temperature gradient, defined as the difference in temperature between the skin surface of the forearm and that of the fingertip (forearm-to-fingertip)
  Other Names: Forearm-to-fingertip temperature gradient
Diagnostic Test: Vaso-occlusion test — Measurement of endothelial function by a vaso-occlusion test performed by inflating a cuff on the arm to occlude arterial flow for 3 min. Reactive hyperemia on deflation of the cuff is measured by photoplethysmography placed on the index finger, and tissue oxygen saturation (StO2) by near-infrared spectroscopy (NIRS). The amplitude of the reperfusion flow corresponding to the peak of the perfusion index (ΔPI Peak) and the time to reach this peak (time to peak) are the parameters recorded by photoplethysmography. Tissue resaturation rate (rStO2) is the parameter recorded by NIRS.
  Other Names: Reactive hyperemia
Diagnostic Test: Transthoracic echocardiography — The diameter of the left ventricular outflow tract is measured in the tele systolic parasternal long-axis view. The pulsed Doppler flow profile is acquired at the level of the left ventricular chamber in the apical five-chamber view. The time-velocity integral of the aortic flow is then calculated. Left ventricular end-diastolic and end-systolic volumes are also measured using Simpson's method in the 4-cavity monoplane view. Measurements of vena cava diameter and respiratory variability of vena cava diameter provide an estimate of right atrial pressure. These measurements estimate cardiac output and systemic vascular resistance.
Diagnostic Test: Photoplethysmography — The perfusion index (PI) is derived from the signal and represents the ratio between the absorbance or reflectance of pulsatile and non-pulsatile light of the photoplethysmography signal. PI is measured non-invasively using a photoplethysmographic sensor placed on the earlobe or finger.
  Other Names: Perfusion index
Procedure: Transcatheter aortic valve insertion (TAVI) — TAVI is a treatment for aortic valve stenosis. A new valve is inserted with minimally invasive procedure without removing the old, damaged valve.
  Other Names: Transcatheter Aortic Valve Replacement (TAVR)

SUMMARY:
The Physiological Study of Haemodynamic and Microcirculatory Evolution before/after Transcatheter Aortic Valve Replacement (TAVI) aims to investigate the physiological changes induced by the implantation of a prosthetic aortic valve on blood vessels in patients with severe aortic stenosis. The hypothesis of the study is that adaptive microcirculatory phenomena occur during TAVI implantation. The results of preoperative assessment of microcirculatory functional reserve differ according to whether or not organ dysfunction occurs after TAVI. There is a progressive adaptation of the microcirculation to the new cardiovascular load conditions after TAVI. Early features of this adaptation are associated with the occurrence of short- and medium-term complications.

DETAILED DESCRIPTION:
This is a prospective, physiologic, monocentric, pilot cohort study carried out at the University Hospitals of Geneva on the initiative of the investigator. We are investigating the adaptive mechanisms at work in the blood vessels and their potential impact on clinical outcomes in the month following surgery. In addition to the usual perioperative monitoring, patients enrolled in the study will benefit from vascular monitoring, which consists of a series of additional non-invasive and painless examinations performed before, a few hours after and on the day after surgery. The clinical outcome of the aortic valve implantation will be monitored by a questionnaire on the day after the procedure, a 6-minute walk test during the usual consultation with the cardiologist on the 6th day after the procedure, and a review of patient health events one month after the valve implantation.

ELIGIBILITY:
Inclusion Criteria:

* All major patients undergoing a femoral TAVI procedure for severe aortic stenosis,

Exclusion Criteria:

* Non-femoral approach for TAVI implantation,
* Presence of other concomitant severe valve disease,
* Planned procedure under general anesthesia,
* Anticipated inability to perform a 6-minute walk test post-operatively (physical handicap),
* Heart failure with left ventricular ejection fraction <40%,
* Chronic end-stage renal failure,
* Chronic lung disease with home oxygen therapy,
* Acquired changes in serum VEGF levels: recent myocardial infarction or stroke, recent vascular intervention (< 3 months), active cancer, anti-angiogenic immunotherapy,
* Patients with known or identified cognitive disorders,
* Persons deprived of their liberty, persons under protective supervision,
* Pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Selection from patients with severe aortic stenosis referred to the Geneva tertiary university hospital for minimally invasive procedures.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2024-05-08 (Actual); Primary Completion 2024-06-13 (Actual); Study Completion 2024-07-13 (Actual)

PRIMARY OUTCOMES:
Modification in arterial stiffness in large- and small-caliber arteries | 24 hours
  Change in arterial stiffness of large/small caliber arteries between preoperative and postoperative measurements.
Modification in plasma Vascular Endothelium Growth Factor levels | 24 hours
  Change in plasma Vascular Endothelium Growth Factor levels between preoperative and postoperative measurements.
Modification in skin surface temperature gradient | 24 hours
  Change in skin surface temperature gradient, defined as the difference in temperature between the skin surface of the forearm and that of the fingertip (forearm-to-fingertip)
Modification in reactive hyperemia | 24 hours
  Change in reactive hyperemia induced by vaso-occlusion test measured by peak of the perfusion index (ΔPI Peak), the time to reach the peak (time to peak), and the tissue resaturation rate (rStO2).

SECONDARY OUTCOMES:
Organ dysfunction | 7 days
  Organ dysfunction: Composite including one of the following events:
  * Acute Kidney Injury (KDIGO classification 1 and above),
  * Acute lung injury (measured or estimated arterial oxygen pressure / inspired oxygen fraction ratio <200),
  * Postoperative cardiovascular failure (need for vasopressor or inotropic support for more than 2 hours),
  * Postoperative neurocognitive impairment assessed using the 3D-Confusion Assessment Method
Functional capacity | day 6
  Distance covered in a 6-minute walk test and percentage of predicted distance
Mortality | 30 days
  All causes mortality
Major Adverse Cardiovascular Events (MACE) | 30 days
  Composite:
  * Acute myocardial infarction, unstable angina, postoperative high-sensitivity troponin (≥ 65 ng/L),
  * Stroke (including transient),
  * Death of cardiovascular origin.
Major Adverse Kidney Events (MAKE) | 30 days
  Composite:
  * Dependence on renal replacement therapy,
  * Decrease in glomerular filtration rate to <75% of baseline,
  * All causes mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Karim Bendjelid, Ph.D., Principal Investigator — University Hospital, Geneva
Locations (1):
- Prof Karim Bendjelid, Geneva, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No